CLINICAL TRIAL: NCT01329029
Title: Effect of Roflumilast on Exacerbation Rate in Patients With COPD Treated With Fixed Combinations of LABA and ICS. A 52-week, Randomised Double-blind Trial With Roflumilast 500 µg Versus Placebo. The REACT Trial
Brief Title: Roflumilast in Chronic Obstructive Pulmonary Disease (COPD) Patients Treated With Fixed Combinations of Long-acting β2-agonists (LABA) and Inhaled Glucocorticosteroid (ICS)
Acronym: REACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RO-2455-404-RD; 2010-019685-87 (EudraCT Number); U1111-1141-7422 (Registry Identifier: WHO)
Record Dates: First submitted 2011-03-30; First posted 2011-04-05 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Roflumilast; Daxas
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast (Active Comparator): concomitant medication: fixed combination of long-acting β2-agonist and inhaled glucocorticosteroid
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): concomitant medication: fixed combination of long-acting β2-agonist and inhaled glucocorticosteroid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 µg, once daily
  Arms: Roflumilast
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
The objective of the REACT trial is to investigate the effect of roflumilast 500 μg tablets once daily versus placebo on exacerbation rate and pulmonary function in COPD patients who are concomitantly treated with a fixed combination of long-acting β2-agonists (LABA) and inhaled glucocorticosteroids (ICS). In addition, data on safety and tolerability of roflumilast will be obtained. An additional objective is to further characterize the population pharmacokinetic profile of roflumilast and roflumilast N oxide and to further characterize their pharmacokinetics/pharmacodynamics (PK/PD) relationship in terms of efficacy and relevant safety aspects.

Patients to be included are required to have severe COPD associated with chronic bronchitis and a history of frequent exacerbations and must be concomitantly treated with a fixed combination of LABA and ICS. Two parallel treatment arms (roflumilast 500 μg once daily and placebo) are included.

DETAILED DESCRIPTION:
The drug tested in this study is called Roflumilast. Roflumilast is being developed to treat people who have chronic obstructive pulmonary disease (COPD). This study investigated the effect of roflumilast 500 μg tablets once daily versus placebo on exacerbation rate, pulmonary function, and major adverse cardiovascular events (MACE) in COPD patients who were concomitantly treated with a fixed combination of long-acting beta-agonists (LABA) and inhaled glucocorticosteroids.

The study was targeted to enroll approximately 1934 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Roflumilast 500 μg once daily
* Placebo (dummy inactive pill) - this was a tablet that looked like the study drug but had no active ingredient

Trial treatment was taken in the morning by mouth after breakfast with some water.

The trial consisted of the following periods:

* Single-blind baseline period (4 weeks) during which all patients received placebo.
* Double-blind treatment period (52 weeks) during which patients received either roflumilast or matching placebo.
* Safety follow-up (30 days after end of treatment (Vend) or premature discontinuation date) in case of ongoing Adverse Events at Vend, if necessary.
* Follow-up visit 12 weeks after end of treatment, at Week 64 (VFU), only for patients who completed the trial as scheduled.

This multi-center trial was conducted worldwide. The overall time to participate in this study was up to 64 weeks. Participants made multiple visits to the clinic which included a follow-up visit at week 64.

ELIGIBILITY:
Inclusion Criteria:

* Giving written informed consent
* History of COPD (according to GOLD 2009) for at least 12 months prior to baseline Visit V0 associated with chronic productive cough for 3 months in each of the 2 years prior to baseline visit (with other causes of productive cough excluded)
* Age ≥ 40 years
* Forced expiratory volume after one second (FEV1)/forced vital capacity (FVC) ratio (post-bronchodilator) < 70%
* FEV1 (post-bronchodilator) ≤ 50% of predicted
* At least two documented moderate or severe COPD exacerbations within one year prior to baseline visit
* Patients must be pre-treated with LABA and ICS for at least 12 months before baseline Visit V0. Up to 3 months before baseline Visit V0 free or fixed combinations of LABA and ICS are allowed, including changes in dose, active substances, and brands. In the last 3 months before baseline Visit V0 patients must be pre-treated with fixed combinations of LABA and ICS at a constant dose (maximum approved dosage strength of the combination).
* Former smoker (defined as smoking cessation at least one year ago) or current smoker both with a smoking history of at least 20 pack years

Main Exclusion Criteria:

* Exacerbations not resolved at first baseline visit
* Diagnosis of asthma and/or other relevant lung disease
* Known alpha-1-antitrypsin deficiency
* Other protocol-defined exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1945 (Actual)
Dates: Start 2011-05; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (159):
- Australia (8):
  - Nycomed Investigational Site, Box Hill
  - Nycomed Investigational Site, Clayton
  - Nycomed Investigational Site, Concord
  - Nycomed Investigational site, Daws Park
  - Nycomed Investigational Site, Frankston
  - Nycomed Investigational Site, Heidelberg
  - Nycomed Investigational Site, Parkville
  - Nycomed Investigational Site, Toorak Gardens
- Austria (4):
  - Nycomed Investigational Site, Feldbach
  - Nycomed Investigational Site, Graz
  - Nycomed Investigational Site, Salzburg
  - Nycomed Investigational Site, Vienna
- Belgium (4):
  - Nycomed Investigational Site, Brussels
  - Nycomed Investigational Site, Halen
  - Nycomed Investigational Site, Liège
  - Nycomed Investigational Site, Malmedy
- Brazil (8):
  - Nycomed Investigational Site, Belo Horizonte
  - Nycomed Investigational Site, Botucatu
  - Nycomed Investigational Site, Florianópolis
  - Nycomed Investigational Site, Goiânia
  - Nycomed Investigational Site, Porto Alegre
  - Nycomed Investigational Site, Rio de Janeiro
  - Nycomed Investigational Site, São Paulo
  - Nycomed Investigational Site, Vitória
- Canada (7):
  - Nycomed Investigational Site, Hamilton
  - Nycomed Investigational Site, Kingston
  - Nycomed Investigational Site, Lachine
  - Nycomed Investigational Site, Niagara Falls
  - Nycomed Investigational Site, Richmond Hill
  - Nycomed Investigational Site, Toronto
  - Nycomed Investigational Site, Winnepeg
- Denmark (4):
  - Nycomed Investigational Site, Hellerup
  - Nycomed Investigational Site, Hillerød
  - Nycomed Investigational Site, Hvidovre
  - Nycomed Investigational Site, København NV
- France (5):
  - Nycomed Investigational Site, Férolles-Attilly
  - Nycomed Investigational Site, Nîmes
  - Nycomed Investigational Site, Poitiers
  - Nycomed Investigational Site, Saint-Laurent-du-Var
  - Nycomed Investigational Site, Strasbourg
- Germany (8):
  - Nycomed Investigational Site, Berlin
  - Nycomed Investigational Site, Fürth
  - Nycomed Investigational Site, Großhansdorf
  - Nycomed Investigational Site, Hanover
  - Nycomed Investigational Site, Homburg
  - Nycomed Investigational Site, Koblenz
  - Nycomed Investigational Site, Marburg
  - Nycomed Investigational Site, Rüdersdorf
- Greece (7):
  - Nycomed Investigational Site, Alexandroupoli
  - Nycomed Investigational Site, Athens
  - Nycomed Investigational Site, Heraklion, Crete
  - Nycomed Investigational Site, Kavala
  - Nycomed Investigational Site, Larissa
  - Nycomed Investigational Site, Marousi
  - Nycomed Investigational Site, Thessaloniki
- Hungary (13):
  - Nycomed Investigational Site, Balassagyarmat
  - Nycomed Investigational Site, Budapest
  - Nycomed Investigational Site, Cegléd
  - Nycomed Investigational Site, Csorna
  - Nycomed Investigational Site, Deszk
  - Nycomed Investigational Site, Érd
  - Nycomed Investigational Site, Miskolc
  - Nycomed Investigational Site, Nyíregyháza
  - Nycomed Investigational Site, Pécs
  - Nycomed Investigational Site, Siófok
  - Nycomed Investigational Site, Sopron
  - Nycomed Investigational Site, Szombathely
  - Nycomed Investigational Site, Törökbálint
- Israel (11):
  - Nycomed Investigational Site, Ashkelon
  - Nycomed Investigational Site, Beersheba
  - Nycomed Investigational Site, Haifa
  - Nycomed Investigational Site, Holon
  - Nycomed Investigational Site, Jerusalem
  - Nycomed Investigational Site, Jerusalm
  - Nycomed Investigational Site, Kfar Saba
  - Nycomed Investigational Site, Petah Tikva
  - Nycomed Investigational Site, Rehovot
  - Nycomed Investigational Site, Tel Aviv
  - Nycomed Investigational Site, Tel Litwinsky
- Italy (7):
  - Nycomed Investigational Site, Ferrara
  - Nycomed Investigational Site, Genova
  - Nycomed Investigational Site, Milan
  - Nycomed Investigational Site, Modena
  - Nycomed Investigational Site, Monza
  - Nycomed Investigational Site, Pordenone
  - Nycomed Investigational Site, Roma
- Netherlands (6):
  - Nycomed Investigational Site, 's-Hertogenbosch
  - Nycomed Investigational Site, Amersfoort
  - Nycomed Investigational Site, Arnhem
  - Nycomed Investigational Site, Enschede
  - Nycomed Investigational Site, Heerlen
  - Nycomed Investigational Site, Hoorn
- Poland (12):
  - Nycomed Investigational Site, Bialystok
  - Nycomed Investigational Site, Bydgoszcz
  - Nycomed Investigational Site, Gliwice
  - Nycomed Investigational Site, Katowice
  - Nycomed Investigational Site, Lodz
  - Nycomed Investigational Site, Lublin
  - Nycomed Investigational Site, Oleśnica
  - Nycomed Investigational Site, Ostrów Wielkopolski
  - Nycomed Investigational Site, Tarnów
  - Nycomed Investigational Site, Warsaw
  - Nycomed Investigational Site, Wroclaw
  - Nycomed Investigational Site, Zawadzkie
- Russia (13):
  - Nycomed Investigational Site, Chelyabinsk
  - Nycomed Investigational Site, Kazan'
  - Nycomed Investigational Site, Kemerovo
  - Nycomed Investigational Site, Moscow
  - Nycomed Investigational Site, Nizhny Novgorod
  - Nycomed Investigational Site, Novosibirsk
  - Nycomed Investigational Site, Saint Petersburg
  - Nycomed Investigational Site, Samara
  - Nycomed Investigational Site, Saratov
  - Nycomed Investigational Site, Smolensk
  - Nycomed Investigational Site, Volgograd
  - Nycomed Investigational Site, Vsevolozhsk
  - Nycomed Investigational Site, Yaroslavl
- Slovakia (8):
  - Nycomed Investigational Site, Banská Bystrica
  - Nycomed Investigational Site, Bardejov
  - Nycomed Investigational Site, Bratislava
  - Nycomed Investigational Site, Košice
  - Nycomed Investigational Site, Martin
  - Nycomed Investigational Site, Nitra
  - Nycomed Investigational Site, Nové Zámky
  - Nycomed Investigational Site, Spišská Nová Ves
- South Africa (10):
  - Nycomed Investigational Site, Auckland Park, Johannesburg Gauteng
  - Nycomed Investigational Site, Benoni Gauteng
  - Nycomed Investigational Site, Bloemfontein Free State
  - Nycomed Investigational Site, Cape Town Western Cape
  - Nycomed Investigational Site, Durban Kwazulu-Natal
  - Nycomed Investigational Site, Johannesburg
  - Nycomed Investigational Site, Morningside, Johannesburg Gauteng
  - Nycomed Investigational Site, Thabazimbi Limpopo
  - Nycomed Investigational Site, Umkomaas Kwazulu-Natal
  - Nycomed Investigational Site, Witbank Mpumalanga
- South Korea (5):
  - Nycomed Investigational Site, Anyang
  - Nycomed Investigational Site, Cheongju-si
  - Nycomed Investigational Site, Daegu
  - Nycomed Investigational Site, Seoul
  - Nycomed Investigational Site, Wŏnju
- Spain (7):
  - Nycomed Investigational Site, Barcelona
  - Nycomed Investigational Site, Guadalajara
  - Nycomed Investigational Site, Madrid
  - Nycomed Investigational Site, Pozuelo de Alarcón
  - Nycomed Investigational Site, Santander
  - Nycomed Investigational Site, Terrassa
  - Nycomed Investigational Site, Valencia
- Turkey (Türkiye) (7):
  - Nycomed Investigational Site, Ankara
  - Nycomed Investigational Site, Çanakkale
  - Nycomed Investigational Site, Istanbul
  - Nycomed Investigational Site, Izmir
  - Nycomed Investigational Site, Kocaeli
  - Nycomed Investigational Site, Konya
  - Nycomed Investigational Site, Mersin
- United Kingdom (5):
  - Nycomed Investigational Site, Edinburgh
  - Nycomed Investigational Site, Glasgow
  - Nycomed Investigational Site, Liverpool
  - Nycomed Investigational Site, London
  - Nycomed Investigational Site, Norwich

REFERENCES:
- [Derived] Facius A, Marostica E, Gardiner P, Watz H, Lahu G. Pharmacokinetic and Pharmacodynamic Modelling to Characterize the Tolerability of Alternative Up-Titration Regimens of Roflumilast in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2018 Aug;57(8):1029-1038. doi: 10.1007/s40262-018-0671-4. PMID 29797235
- [Derived] Martinez FJ, Rabe KF, Calverley PMA, Fabbri LM, Sethi S, Pizzichini E, McIvor A, Anzueto A, Alagappan VKT, Siddiqui S, Reisner C, Zetterstrand S, Roman J, Purkayastha D, Bagul N, Rennard SI. Determinants of Response to Roflumilast in Severe Chronic Obstructive Pulmonary Disease. Pooled Analysis of Two Randomized Trials. Am J Respir Crit Care Med. 2018 Nov 15;198(10):1268-1278. doi: 10.1164/rccm.201712-2493OC. PMID 29763572
- [Derived] Rabe KF, Calverley PMA, Martinez FJ, Fabbri LM. Effect of roflumilast in patients with severe COPD and a history of hospitalisation. Eur Respir J. 2017 Jul 5;50(1):1700158. doi: 10.1183/13993003.00158-2017. Print 2017 Jul. No abstract available. PMID 28679611
- [Derived] Martinez FJ, Calverley PM, Goehring UM, Brose M, Fabbri LM, Rabe KF. Effect of roflumilast on exacerbations in patients with severe chronic obstructive pulmonary disease uncontrolled by combination therapy (REACT): a multicentre randomised controlled trial. Lancet. 2015 Mar 7;385(9971):857-66. doi: 10.1016/S0140-6736(14)62410-7. Epub 2015 Feb 13. PMID 25684586
- [Derived] Calverley PM, Martinez FJ, Fabbri LM, Goehring UM, Rabe KF. Does roflumilast decrease exacerbations in severe COPD patients not controlled by inhaled combination therapy? The REACT study protocol. Int J Chron Obstruct Pulmon Dis. 2012;7:375-82. doi: 10.2147/COPD.S31100. Epub 2012 Jun 20. PMID 22791991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 203 investigative sites in Australia, Austria, Belgium, Brazil, Canada, Denmark, France, Germany, Greece, Hungary, Israel, Italy, Korea (Republic of), Netherlands, Poland, Russia, Slovak Republic, South Africa, Spain, Turkey and United Kingdom from 28 May 2011 to 27 May 2014.
Pre-assignment Details: Participants with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) entered a 4 week baseline period during which all patients received placebo then were enrolled equally in 1 of 2 treatment groups, once a day placebo or roflumilast 500 µg.
Groups:
- Roflumilast 500 µg: Roflumilast 500 µg tablet, orally, once daily for 52 weeks. Background therapy concomitant medication: fixed combination of long-acting β2-agonist and inhaled glucocorticosteroid.
- Placebo: Placebo-matching roflumilast tablet, orally, once daily for 52 weeks. Background therapy concomitant medication: fixed combination of long-acting β2-agonist and inhaled glucocorticosteroid.
Period: Overall Study
Arm/Group | Roflumilast 500 µg | Placebo
Started | 973 | 972
Full Analysis Set (FAS) | 969 | 966
Safety Population | 968 | 967
Completed | 704 | 780
Not Completed | 269 | 192
Not completed — Withdrawal by Subject | 117 | 87
Not completed — Adverse Event | 82 | 29
Not completed — Death | 16 | 19
Not completed — Other | 14 | 20
Not completed — COPD Exacerbation | 11 | 18
Not completed — Physician Decision | 16 | 13
Not completed — Lost to Follow-up | 8 | 5
Not completed — Met Pre-defined Discontinuation Criteria | 5 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all randomised participants who took at least 1 dose of investigational medicinal product (IMP) after randomisation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast 500 µg | Placebo | Total
Number analyzed (Participants) | 969 | 966 | 1935
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (8.38) | 64.7 (8.37) | 64.7 (8.37)
Age, Customized [Number; unit: participants]
  ≤ 65 years | 527 | 542 | 1069
  > 65 years | 442 | 424 | 866
Gender [Count of Participants; unit: Participants]
  Female | 251 | 241 | 492
  Male | 718 | 725 | 1443
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 20 | 16 | 36
  Black or African American | 6 | 5 | 11
  White | 940 | 943 | 1883
  Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Australia | 9 | 16 | 25
  Austria | 11 | 3 | 14
  Belgium | 19 | 18 | 37
  Brazil | 42 | 38 | 80
  Canada | 14 | 12 | 26
  Denmark | 15 | 19 | 34
  France | 16 | 13 | 29
  Germany | 70 | 63 | 133
  Greece | 38 | 30 | 68
  Hungary | 111 | 125 | 236
  Israel | 114 | 126 | 240
  Italy | 64 | 51 | 115
  Korea, Republic Of | 11 | 7 | 18
  Netherlands | 11 | 8 | 19
  Poland | 88 | 88 | 176
  Russian Federation | 177 | 181 | 358
  Slovakia | 25 | 33 | 58
  South Africa | 23 | 30 | 53
  Spain | 37 | 33 | 70
  Turkey | 52 | 44 | 96
  United Kingdom | 22 | 28 | 50
Height [Mean (Standard Deviation); unit: cm] | 168.20 (8.652) | 168.33 (8.198) | 168.26 (8.427)
Weight [Mean (Standard Deviation); unit: kg] | 75.07 (17.275) | 75.60 (17.238) | 75.33 (17.254)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.45 (5.474) | 26.58 (5.359) | 26.52 (5.416)
Chronic Obstructive Pulmonary Disease (COPD) Severity [Number; unit: participants] — COPD severity was classified according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guideline (2009) as: - Very severe COPD: baseline post-bronchodilator FEV1 %predicted < 30% - Severe COPD: baseline post-bronchodilator FEV1 %predicted ≥ 30% to < 50% - Moderate COPD: baseline post-bronchodilator FEV1 %predicted ≥ 50% to < 80% - Mild COPD: baseline post-bronchodilator FEV1 %predicted ≥ 80%.
  participants
    Mild | 2 | 0 | 2
    Moderate | 18 | 16 | 34
    Severe | 658 | 677 | 1335
    Very Severe | 291 | 273 | 564
COPD Disease Characteristics [Number; unit: participants]
  Pure emphysema | 4 | 2 | 6
  Predominantly chronic bronchitis | 338 | 330 | 668
  Combined emphysema and chronic bronchitis | 626 | 634 | 1260
  Missing | 1 | 0 | 1
Global Initiative for Chronic Obstructive Lung Disease (GOLD) Patient Group [Number; unit: participants]
  A : low risk, less symptoms | 0 | 0 | 0
  B: low risk, more symptoms | 0 | 0 | 0
  C: high risk, less symptoms | 62 | 57 | 119
  D: high risk, more symptoms | 905 | 907 | 1812
  Missing | 2 | 2 | 4
Smoking Status [Number; unit: participants]
  Current smoker | 411 | 432 | 843
  Former smoker | 558 | 534 | 1092
  Nonsmoker | 0 | 0 | 0
Cigarette Pack Years [Mean (Standard Deviation); unit: pack years] — Pack Years = (packs smoked per day) * (years as a smoker)
  pack years | 47.6 (24.55) | 47.6 (23.56) | 47.6 (24.6)
Pre-bronchodilator Forced Expiratory Volume in the First Second (FEV1) [Mean (Standard Deviation); unit: Liters] — Number of participants for whom pre-bronchodilator FEV1 data was available was 938 and 937 in each treatment arm, respectively.
  Liters | 0.999 (0.3149) | 1.016 (0.3209) | 1.008 (0.3180)
Post-bronchodilator FEV1 [Mean (Standard Deviation); unit: Liters] | 1.066 (0.3317) | 1.078 (0.3244) | 1.072 (0.3280)
Pre-bronchodilator FEV1 Predicted [Mean (Standard Deviation); unit: percent of predicted] — Number of participants for whom pre-bronchodilator FEV1 data was available was 938 and 933 in each treatment arm, respectively.
  percent of predicted | 33.259 (9.0781) | 33.562 (9.0043) | 33.411 (9.0402)
Post-bronchodilator FEV1 Predicted [Mean (Standard Deviation); unit: percent predicted] | 35.392 (9.2484) | 35.532 (8.7573) | 35.462 (9.0045)
FEV1 Reversibility % Increase [Mean (Standard Deviation); unit: percent reversibility] — FEV reversibility (%) = (post-bronchodilator FEV minus pre-bronchodilator FEV) / pre-bronchodilator FEV * 100. Number of participants for whom FEV1 reversibility % increase data was available was 912 and 915 in each treatment arm, respectively.
  percent reversibility | 7.465 (11.2559) | 7.383 (12.0752) | 7.424 (11.6703)
FEV1 Reversibility Increase [Mean (Standard Deviation); unit: mL] — Number of participants for whom FEV1 reversibility increase data was available was 912 and 915 in each treatment arm, respectively.
  mL | 65.2 (108.72) | 65.4 (121.55) | 65.3 (115.29)
Post-bronchodilator FEV1/Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: FEV1/FVC percent] — Calculated as FEV1/FVC * 100
  FEV1/FVC percent | 40.2 (10.81) | 40.1 (10.26) | 40.1 (10.54)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate or Severe COPD Exacerbations Per Patient Per Year
Description: A COPD exacerbation is an event in the natural course of the disease characterized by a worsening in the patient's baseline dyspnoea, cough, and/or sputum production beyond day to day variability sufficient to warrant a change in management. COPD exacerbations were categorized as follows: Severe=Requiring hospitalization and/or leading to death; Moderate=Requiring oral or parenteral glucocorticosteroid therapy. The defined number of days a patient was in the trial was divided by 365.25, in order to express the duration as a fraction of 1 year.
Time Frame: 52 weeks
Population: Participants from the Intent-to treat population, all randomized participants who received at least 1 dose of study drug analyzed by the treatment for which they were randomized, with data available for analysis.
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient per year
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
exacerbations per patient per year | 0.805 [0.724 to 0.895] | 0.927 [0.843 to 1.020]
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.0529, Generalized Linear Regression — Level of significance: 5% 2-sided; Poisson regression model (estimates of exacerbation rates using time in trial as model offset); Rate ratio = 0.868, 95% CI 2-sided [0.753 to 1.002], Standard Error of Mean 0.0633 — A rate ratio of < 1 represents a favourable outcome for the test treatment

2. Secondary Outcome: Change From Baseline in Post-Bronchodilator Forced Expiratory Volume in the First Second (FEV1)
Description: Pulmonary function testing was performed using centralised spirometry. FEV1 is the maximum amount of air that can be forcefully exhaled in one second. Least-squares means is from Analysis of Covariance (ANCOVA) including treatment by time interaction. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 928 | 941
liters | 0.052 (0.0064) | -0.004 (0.0062)
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Analysis of Covariance (ANCOVA) including treatment by time interaction; LS Mean difference = 0.056, 95% CI 2-sided [0.038 to 0.073], Standard Error of Mean 0.0089

3. Secondary Outcome: Rate of Severe COPD Exacerbations Per Patient Per Year
Description: A COPD exacerbation is an event in the natural course of the disease characterized by a worsening in the patient's baseline dyspnoea, cough, and/or sputum production beyond day to day variability sufficient to warrant a change in management. Severe COPD exacerbations were categorized as requiring hospitalization and/or leading to death. The defined number of days a patient was in the trial was divided by 365.25, in order to express the duration as a fraction of 1 year.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient per year
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
exacerbations per patient per year | 0.239 [0.201 to 0.283] | 0.315 [0.270 to 0.368]
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.0175, Generalized Linear Regression; Analyzed using a negative binomial regression model excluding a correction for overdispersion; Rate ratio = 0.757, 95% CI 2-sided [0.601 to 0.952], Standard Error of Mean 0.0889 — A rate ratio of < 1 represents a favourable outcome for the test treatment

4. Secondary Outcome: Rate of COPD Exacerbations Per Patient Per Year All Categories
Description: as for outcome 1
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient per year
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
exacerbations per patient per year
  Moderate | 0.574 [0.508 to 0.648] | 0.627 [0.561 to 0.702]
  Mild, Moderate or Severe | 3.078 [2.723 to 3.479] | 3.879 [3.492 to 4.310]
  Leading to Hospitalisation | 0.238 [0.200 to 0.283] | 0.313 [0.268 to 0.365]
  Glucocorticosteroids and/or Antibiotics treatment | 0.794 [0.716 to 0.88] | 0.929 [0.847 to 1.019]
  Moderate or Severe and/or treated with Antibiotics | 1.012 [0.922 to 1.110] | 1.210 [1.115 to 1.313]
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Moderate COPD Exacerbations; Test type: Superiority or Other; p = 0.2875, Generalized Linear Regression — Level of significance: 5% 2-sided; Poisson regression model (estimates of exacerbation rates using time in trial as model offset); Rate ratio = 0.914, 95% CI 2-sided [0.775 to 1.078], Standard Error of Mean 0.0771 — A rate ratio of < 1 represents a favourable outcome for the test treatment
Statistical Analysis 2: Comparison: Roflumilast 500 µg vs Placebo; Mild, Moderate or Severe COPD Exacerbations; Test type: Superiority or Other; p = 0.0050, Generalized Linear Regression — Level of significance: 5% 2-sided; Poisson regression model (estimates of exacerbation rates using time in trial as model offset); Rate Ratio = 0.794, 95% CI 2-sided [0.675 to 0.933], Standard Error of Mean 0.0654 — A rate ratio of < 1 represents a favourable outcome for the test treatment
Statistical Analysis 3: Comparison: Roflumilast 500 µg vs Placebo; COPD Exacerbations treated with Glucocorticosteroids and/or Antibiotics; Test type: Superiority or Other; p = 0.0262, Generalized Linear Regression — Level of significance: 5% 2-sided; Poisson regression model (estimates of exacerbation rates using time in trial as model offset); Rate ratio = 0.854, 95% CI 2-sided [0.744 to 0.982], Standard Error of Mean 0.0605 — A rate ratio of < 1 represents a favourable outcome for the test treatment
Statistical Analysis 4: Comparison: Roflumilast 500 µg vs Placebo; Moderate or Severe COPD Exacerbations and/or treated with Antibiotics; Test type: Superiority or Other; p = 0.0047, Generalized Linear Regression — Level of significance: 5% 2-sided; Poisson regression model (estimates of exacerbation rates using time in trial as model offset); Rate ratio = 0.837, 95% CI 2-sided [0.739 to 0.947], Standard Error of Mean 0.0528 — A rate ratio of < 1 represents a favourable outcome for the test treatment
Statistical Analysis 5: Comparison: Roflumilast 500 µg vs Placebo; Leading to Hospitalisation; Test type: Superiority or Other; p = 0.0209, Generalized Linear Regression — Level of significance: 5% 2-sided; Negative binomial regression model (estimates of exacerbation rates); Rate ratio = 0.761, 95% CI 2-sided [0.604 to 0.960], Standard Error of Mean 0.0899 — A rate ratio of < 1 represents a favourable outcome for the test treatment

5. Secondary Outcome: Percentage of Participants Experiencing at Least 1 COPD Exacerbation
Description: A COPD exacerbation is an event in the natural course of the disease characterized by a worsening in the patient's baseline dyspnoea, cough, and/or sputum production beyond day to day variability sufficient to warrant a change in management.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
percentage of participants | 55.2 | 60.5

6. Secondary Outcome: Time to First COPD Exacerbation All Categories
Description: Time to event was calculated as date of onset of event - date of first intake of double-blind study drug + 1 day for all events: mild, moderate or severe. A COPD exacerbation is an event in the natural course of the disease characterized by a worsening in the patient's baseline dyspnoea, cough, and/or sputum production beyond day to day variability sufficient to warrant a change in management.
Time Frame: 52 Weeks
Population: Participants from the Intent-to treat population, all randomized participants who received at least 1 dose of study drug analyzed by the treatment for which they were randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | 218.0 [189.0 to 259.0] | 180.0 [147.0 to 200.0]
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.1461, Cox proportional hazards model — Level of significance: 5% 2-sided; Hazard Ratio (HR) = 0.917, 95% CI 2-sided [0.815 to 1.031], Standard Error of Mean 0.0549 — A hazards ratio of < 1 represents a lower hazard for the test treatment

7. Secondary Outcome: Time to Second Moderate or Severe COPD Exacerbation
Description: Time to event was calculated as date of onset of event - date of first intake of double-blind study drug + 1 day for events: moderate or severe. A COPD exacerbation is an event in the natural course of the disease characterized by a worsening in the patient's baseline dyspnoea, cough, and/or sputum production beyond day to day variability sufficient to warrant a change in management. COPD exacerbations were categorized as Severe: Requiring hospitalization and/or leading to death; Moderate: Requiring oral or parenteral glucocorticosteroid therapy.
Time Frame: 52 Weeks (some participants extended treatment beyond 52 Weeks and are included in the analysis)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | 421.0 [413.0 to NA] — 95% confidence interval upper limit not estimated. | NA [NA to NA] — Parameters not estimated-data did not reach the median.
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.0270, Wei-Lin-Weissfeld Method — Level of significance: 5% 2-sided; Hazard Ratio (HR) = 0.790, 95% CI 2-sided [0.641 to 0.974], Standard Error of Mean 0.0842 — A hazard ratio of <1 represents a favourable outcome for the test treatment

8. Secondary Outcome: Time to Third Moderate or Severe COPD Exacerbation
Description: as for outcome 7
Time Frame: 52 Weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | NA [NA to NA] — Parameters not estimated-data did not reach the median. | NA [NA to NA] — Parameters not estimated-data did not reach the median.
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.0731, Wei-Lin-Weissfeld Method — Level of significance: 5% 2-sided; Hazard Ratio (HR) = 0.749, 95% CI 2-sided [0.546 to 1.027], Standard Error of Mean 0.1209 — A hazard ratio of <1 represents a favourable outcome for the test treatment

9. Secondary Outcome: Number of Patients Needed to Treat to Avoid 1 Moderate or Severe COPD Exacerbation Derived From Exacerbation Per Patient Per Year
Description: The number needed to treat (NNT) analysis is a simple, concise method to quantify directly the benefits that alternative treatment options have on disease outcomes in terms of the number of patients who need to be treated before a benefit is observed. Risk reduction: Rate(Placebo)- Rate (Roflumilast 500 μg), Number needed to treat for benefit (NNTB): 1/(Risk reduction). A COPD exacerbation is an event in the natural course of the disease characterized by a worsening in the patient's baseline dyspnoea, cough, and/or sputum production beyond day to day variability sufficient to warrant a change in management. COPD exacerbations were categorized as Severe: Requiring hospitalization and/or leading to death; Moderate: Requiring oral or parenteral glucocorticosteroid therapy.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
participants | 0.805 | 0.927
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; NNTB = 9, 95% CI 2-sided [4 to 31]

10. Secondary Outcome: Number of Moderate or Severe COPD Exacerbation Days
Description: A COPD exacerbation is an event in the natural course of the disease characterized by a worsening in the patient's baseline dyspnoea, cough, and/or sputum production beyond day to day variability sufficient to warrant a change in management. The number of exacerbation days per patient is the sum of durations (stop date of exacerbation - start date of exacerbation + 1) of all exacerbations within the category.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 380 | 432
days | 26.9 (23.09) | 30.9 (29.49)

11. Secondary Outcome: Duration of Moderate or Severe COPD Exacerbations Per Participant
Description: as for outcome 5
Time Frame: 52 Weeks
Population: Participants from the Intent-to treat population, all randomized participants who received at least 1 dose of study drug analyzed by the treatment for which they were randomized, with data available for analysis. n in each of the categories is the number of participants with exacerbations.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 380 | 432
days | 15.9 (10.59) | 16.6 (14.49)

12. Secondary Outcome: Change From Baseline in Post-Bronchodilator Forced Vital Capacity (FVC)
Description: Forced vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Least-squares means was from ANCOVA including treatment by time interaction. A positive change from Baseline indicates improvement.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 928 | 941
liters | 0.036 (0.0114) | -0.057 (0.0111)
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p < 0.0001, Repeated measurement model — Level of significance: 5% 2-sided; Unstructured covariance structure and restricted maximum likelihood (REML); Least Square Mean Difference = 0.092, 95% CI 2-sided [0.061 to 0.124], Standard Error of Mean 0.0159

13. Secondary Outcome: Change From Baseline in Post-Bronchodilator Forced Expiratory Flow at 25% to 75% of Vital Capacity (FEF25-75%)
Description: Forced expiratory flow 25-75% (FEF25-75%) is the flow (or speed) of air coming out of the lung during the middle half of a forced expiration. Pulmonary function testing was performed using centralized spirometry. Least-squares means was from ANCOVA including treatment by time interaction. A positive change from Baseline indicates improvement.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 928 | 941
liters/second | 0.035 (0.0044) | 0.009 (0.0043)
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p < 0.0001, Repeated measurement model — Level of significance: 5% 2-sided; Unstructured covariance structure and REML; Least Square Mean Difference = 0.025, 95% CI 2-sided [0.013 to 0.038], Standard Error of Mean 0.0062

14. Secondary Outcome: Change From Baseline in Post-Bronchodilator Forced Expiratory Volume in the First 6 Seconds (FEV6)
Description: FEV6 is the amount of air which can be forcibly exhaled from the lungs in the first six seconds of a forced exhalation. Pulmonary function testing was performed using centralized spirometry. A positive change from Baseline indicates improvement.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 924 | 937
liters | 0.061 (0.0093) | -0.033 (0.0091)
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p < 0.0001, Repeated measurement model — Level of significance: 5% 2-sided; Unstructured covariance structure and REML; Least Square Mean Difference = 0.094, 95% CI 2-sided [0.069 to 0.120], Standard Error of Mean 0.0131

15. Secondary Outcome: Change From Baseline in Post-Bronchodilator FEV1/FVC
Description: The FEV1/FVC ratio represents the percentage of vital capacity expelled from the lungs during the first second of a forced exhalation. Pulmonary function testing was performed using centralized spirometry. A positive change from Baseline indicates improvement.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 701 | 780
percent | 1.170 (7.0339) | 0.580 (6.8405)

16. Secondary Outcome: Change From Baseline in Use of Rescue Medication From Daily Diary
Description: Salbutamol metered dose inhaler was available as rescue medication during the study. The participant recorded the use of rescue medication in a daily diary. A negative change from Baseline indicates an improvement.
Time Frame: Baseline and Week 52
Population: Participants from the Intent-to treat population, all randomized participants who received at least 1 dose of study drug analyzed by the treatment for which they were randomized, with data included in the repeated measurements analysis.
Measure: Least Squares Mean (Standard Error); unit: puffs per day
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 848 | 896
puffs per day | -0.109 (0.0676) | 0.173 (0.0654)
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.0027, Repeated measurement model — Level of significance: 5% 2-sided; Compound symmetry covariance structure and REML; Least Square Mean Difference = -0.283, 95% CI 2-sided [-0.467 to -0.098], Standard Error of Mean 0.0941

17. Secondary Outcome: Change From Baseline in COPD Symptom Score From Daily Diary
Description: Participants recorded COPD symptoms cough and sputum production in a daily diary. Cough was assessed using a 4-point scale where 0=No cough to 3=severe cough and sputum was assessed using a 4-point scale where 0=no sputum production to 3=severe sputum production. Least-squares means from ANCOVA including treatment by time interaction. A negative change from Baseline indicates improvement. Total symptom score is the sum of cough and sputum scores, ranging from 0 (best possible outcome) to 6 (worst possible outcome).
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 897 | 932
score on a scale | -0.412 (0.0315) | -0.398 (0.0306)
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.7392, Repeated measurement model — Level of significance: 5% 2-sided; Compound symmetry covariance structure and REML; Least Square Mean Difference = -0.015, 95% CI 2-sided [-0.101 to 0.071], Standard Error of Mean 0.0439

18. Secondary Outcome: Percentage of Symptom-Free Days
Description: Symptoms of COPD (cough, sputum) were recorded in a daily diary. The percentage of days without symptoms is reported.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
percentage of days | 7.09 (17.119) | 6.88 (16.185)

19. Secondary Outcome: Percentage of Rescue Medication-Free Days
Description: Participants recorded their use of rescue medication in a daily diary. The percentage of days without rescue medication use.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
percentage of days | 23.25 (33.734) | 22.77 (33.141)

20. Secondary Outcome: Change From Baseline in COPD Assessment Test (CAT) Total Score
Description: Participants completed the CAT questionnaire at Baseline and after 52 Weeks of Treatment. The CAT questionnaire measures the impact of COPD on wellbeing and daily life. Participants answer 8 questions on a scale from 0 (best) to 5 (worst). The total score ranges from 0 to 40 with higher scores indicating more impact. A negative change from Baseline indicates improvement. Least-squares means from ANCOVA including treatment by time interaction.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 924 | 940
score on a scale | -1.270 (0.1556) | -0.985 (0.1518)
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.1909, Repeated measurement model — Level of significance: 5% 2-sided; Unstructured covariance structure and REML; Least Square Mean Difference = -0.285, 95% CI 2-sided [-0.711 to 0.142], Standard Error of Mean 0.2175

21. Secondary Outcome: Percentage of Participants With Improvement in CAT
Description: Participants completed the CAT questionnaire at Baseline and after 52 Weeks of treatment. The CAT questionnaire measures the impact of COPD on wellbeing and daily life. Participants answer 8 questions on a scale from 0 (best) to 5 (worst). The total score ranges from 0 to 40 with higher scores indicating more impact. Improvement was defined as a CAT Total Score reduction from Baseline > 1.6.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
percentage of participants | 71.2 | 72.5

22. Secondary Outcome: Time to Mortality Due to Any Reason During the Treatment Period Score
Description: Time to event will be calculated as date of onset of event - date of first intake of double-blind study drug + 1 day.
Time Frame: 52 Weeks (some participants extended treatment beyond 52 Weeks and are included in the analysis)
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | NA [44 to 381] — Data did not reach the median. | NA [21 to 293] — Data did not reach the median.
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.9414, Cox-proportional hazards model — Level of significance: 5% 2-sided; Hazard Ratio (HR) = 1.025, 95% CI 2-sided [0.528 to 1.990], Standard Error of Mean 0.3468 — A hazards ratio of < 1 represents a lower hazard for the test treatment

23. Secondary Outcome: Time to Mortality Due to COPD Exacerbation During the Treatment Period
Description: Time to event will be calculated as date of onset of event - date of first intake of double-blind study drug + 1 day.
Time Frame: 52 Weeks
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | NA [44 to 322] — Data did not reach the median. | NA [25 to 293] — Data did not reach the median.
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.8876, Cox-proportional hazards model; Level of significance: 5% 2-sided; Hazard Ratio (HR) = 1.078, 95% CI 2-sided [0.378 to 3.075], Standard Error of Mean 0.5765 — A hazards ratio of < 1 represents a lower hazard for the test treatment

24. Secondary Outcome: Time to Withdrawal During the Treatment Period
Description: Time to event will be calculated as date of onset of event - date of first intake of double-blind study drug + 1 day.
Time Frame: 52 Weeks (some participants extended treatment beyond 52 Weeks and are included in the analysis)
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | 420.0 [5 to 428] | 444.0 [1 to 444]
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p < 0.0001, Cox-proportional hazards model; Level of significance: 5% 2-sided; Hazard Ratio (HR) = 1.529, 95% CI 2-sided [1.268 to 1.845], Standard Error of Mean 0.1463 — A hazards ratio of < 1 represents a lower hazard for the test treatment

25. Secondary Outcome: Time to Withdrawal Due to COPD Exacerbation During the Treatment Period
Description: Time to event will be calculated as date of onset of event - date of first intake of double-blind study drug + 1 day.
Time Frame: 52 Weeks (some participants extended treatment beyond 52 Weeks and are included in the analysis)
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | NA [25 to 371] — Data did not reach the median. | NA [12 to 319] — Data did not reach the median.
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.3477, Cox-proportional hazards model — Level of significance: 5% 2-sided; Hazard Ratio (HR) = 0.695, 95% CI 2-sided [0.326 to 1.484], Standard Error of Mean 0.2691 — A hazards ratio of < 1 represents a lower hazard for the test treatment

26. Secondary Outcome: Percentage of Participants With Major Adverse Cardiovascular Event (MACE) During the Treatment Period
Description: Composite MACE is a combined endpoint (cardiovascular death [including death due to undetermined cause], nonfatal myocardial infarction, and nonfatal stroke).
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
percentage of participants | 1.7 | 1.7

27. Secondary Outcome: Time to First Major Adverse Cardiovascular Event (MACE) During the Treatment Period
Description: Composite MACE is a combined endpoint(cardiovascular death [including death due to undetermined cause], nonfatal myocardial infarction, and nonfatal stroke). Time to event was calculated as date of onset of event - date of first intake of double-blind study drug + 1 day.
Time Frame: 52 Weeks (some participants extended treatment beyond 52 Weeks and are included in the analysis)
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | NA [52 to 415] — Data did not reach the median. | NA [50 to 365] — Data did not reach the median.
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.8208, Cox-proportional hazards model — Level of significance: 5% 2-sided; Hazard Ratio (HR) = 1.083, 95% CI 2-sided [0.542 to 2.167], Standard Error of Mean 0.3832 — A hazards ratio of < 1 represents a lower hazard for the test treatment

28. Secondary Outcome: Percentage of Participant With All-Cause Hospitalisation During the Treatment Period
Description: Percentage of patients with at least one hospital admission due to any cause.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
percentage of participants | 24.9 | 29.3

29. Secondary Outcome: Time to First Hospitalisation Due to Any Cause During the Treatment Period
Description: Time to event will be calculated as date of onset of event - date of first intake of double-blind study drug + 1 day.
Time Frame: 52 Weeks (some participants extended treatment beyond 52 Weeks and are included in the analysis)
Population: Participants from the Intent-to treat population, all randomized participants who received at least 1 dose of study drug analyzed by the treatment for which they were randomized, with events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | 400.0 [387.0 to 415.0] | 408.0 [391.0 to 420.0]
Statistical Analysis 1: Comparison: Roflumilast 500 µg vs Placebo; Test type: Superiority or Other; p = 0.7943, Cox-proportional hazards model — Level of significance: 5% 2-sided; Hazard Ratio (HR) = 0.977, 95% CI 2-sided [0.821 to 1.162], Standard Error of Mean 0.0865

30. Secondary Outcome: Time to Trial Withdrawal Due to an Adverse Event
Description: Time to event will be calculated as date of onset of event - date of first intake of double-blind study drug + 1 day.
Time Frame: 52 Weeks (some participants extended treatment beyond 52 Weeks and are included in the analysis)
Population: as for outcome 29
Measure: Median (Full Range); unit: days
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 969 | 966
days | NA [7 to 420] — Data did not reach the median. | NA [13 to 444] — Data did not reach the median.

31. Secondary Outcome: Percentage of Participants Who Experienced at Least 1 Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: 52 Weeks
Population: Safety Population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 968 | 967
percentage of participants | 66.9 | 59.2

32. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Square Means was from an ANCOVA model including Last Observation Carried Forward (LOCF).
Time Frame: Baseline and Week 52
Population: Participants from the Safety Population, all randomized participants who received at least one dose of study drug, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 938 | 944
kilogram (kg) | -2.66 (0.130) | -0.14 (0.130)

33. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Body mass index (BMI) is a measure of body fat based on height and weight. Least Square Means was from an ANCOVA model including LOCF.
Time Frame: Baseline and Week 52
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Roflumilast 500 µg | Placebo
Number analyzed (Participants) | 938 | 944
kg/m^2 | -0.94 (0.046) | -0.04 (0.046)

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Safety Population included all randomized participants who received at least one dose of study drug.
Arm/Group | Roflumilast 500 µg | Placebo
Serious Adverse Events (participants affected / at risk) | 249/968 | 285/967
Other Adverse Events (participants affected / at risk) | 228/968 | 114/967
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast 500 µg (N=968) | Placebo (N=967)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 1 | 5
Angina unstable (Cardiac disorders) | 0 | 2
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 6
Atrial flutter (Cardiac disorders) | 2 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 5
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 2
Cardiogenic shock (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 0 | 2
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 5
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Accessory auricle (Congenital, familial and genetic disorders) | 1 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2
Thyrotoxic crisis (Endocrine disorders) | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Eye haemorrhage (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 3 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 3 | 2
Drug ineffective (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 3
Pain (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Bronchopneumonia (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Extradural abscess (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 | 7
Laryngitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Parotid abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 33 | 37
Pneumonia moraxella (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection viral (Infections and infestations) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Transplant evaluation (Investigations) | 1 | 0
Weight decreased (Investigations) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Eyelid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid sinus syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal mass (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 144 | 184
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Alcohol detoxification (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 2
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Leriche syndrome (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast 500 µg (N=968) | Placebo (N=967)
Diarrhoea (Gastrointestinal disorders) | 97 | 33
Nausea (Gastrointestinal disorders) | 55 | 15
Nasopharyngitis (Infections and infestations) | 52 | 52
Weight decreased (Investigations) | 84 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.